CLINICAL TRIAL: NCT02024594
Title: Comparison of Effect of Nitrous Oxide-Oxygen Conscious Sedation and Cognitive-behavioral Therapy on Children's Anxiety in Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fatemeh Mazhari, principle investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 88311
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Clinical Anxiety; Clinical Cooperation
Keywords: Nitrous Oxide-Oxygen conscious sedation; Cognitive Behavioral Therapy; Children, Preschool; dental anxiety; Patient Cooperation
MeSH Terms: conditions — Patient Compliance | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nitrous Oxide-Oxygen (Experimental): Children in this group were sedated by rapid induction method by means of Nitrous Oxide-Oxygen gas.
  Interventions: Drug: Nitrous Oxide-Oxygen conscious sedation
- cognitive-behavioral therapy (Experimental): Children in this group were asked to come to playroom before entering operation room. Modeling , Benson relaxation and positive self-talking were instructed to them.
  Interventions: Behavioral: cognitive-behavioral therapy
- control (No Intervention): No intervention

INTERVENTIONS:
Drug: Nitrous Oxide-Oxygen conscious sedation
  Arms: Nitrous Oxide-Oxygen
Behavioral: cognitive-behavioral therapy
  Arms: cognitive-behavioral therapy

SUMMARY:
Visiting anxious and fearful children is an inevitable prospect of the daily work of every dentist who treats pediatric patients. Dentists have been using a wide variety of non-pharmacological and some pharmacologic techniques to assist them in the management of children with anxiety. One strategy which seems promising for pain control in stressful medical situations is teaching the child to use behavioral and cognitive coping skills or a combination of both techniques. An alternative technique to non-pharmacologic approaches in children being anxious and lacking in cooperative ability is sedative technique such as nitrous oxide conscious sedation. As there is lack of studies comparing conscious sedation and combinations of cognitive-behavioral strategies in eliminating children's uncooperative behaviors and dental anxiety, the aim of this study was to compare the effectiveness of inhalation sedation with Nitrous Oxide-Oxygen conscious sedation and cognitive-behavioral therapy to reduce dental anxiety in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Age between3 to 6.5 year of old
* Presence of moderate to severe dental anxiety
* Parents' acceptance to cooperate in sampling process and 2 sessions of dental treatment
* Presence of at least one mandibular primary molar needed pulp treatment
* positive dental history

Exclusion Criteria:

* current episodes of medications or drug therapy
* systemic or congenital disorders
* mental retardation

Ages: 36 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
change from baseline in Clinical Anxiety and Cooperation scales. | baseline and 1 week
  The anxiety and cooperation differences between the two dental visits (second visits were done after 1 week) were compared within the three groups.